CLINICAL TRIAL: NCT03713905
Title: A Phase I Study to Investigate the Safety, Tolerability, Pharmacokinetics and Antitumor Activities of the Recombinant Human Anti-PD-1 Monoclonal Antibody for Subjects With Advanced Solid Tumors
Brief Title: Study of Recombinant Human Anti-PD-1 Monoclonal Antibody for Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Gloria Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YH-S001-01
Record Dates: First submitted 2018-09-25; First posted 2018-10-22 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — zimberelimab

STUDY DESIGN:
Intervention Model Description: 1 mg per kg, Q2W; 4 mg per kg, Q2W; 10 mg per kg, Q2W; 240 mg fixed dose, Q2W
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GLS-010 (Experimental): Use Full-human anti-pd-1 monoclonal antibodies for treatment
  Interventions: Drug: GLS-010

INTERVENTIONS:
Drug: GLS-010 — Recombinant Human Anti-PD-1 Monoclonal Antibody
  Other Names: Recombinant Human Anti-PD-1 Monoclonal Antibody

SUMMARY:
To investigate the safety and tolerability of GLS-010 in subjects with advanced solid tumors (mainly gastric cancer, esophageal cancer).

To investigate the preliminary relationship between the expression of the ligand of PD-1 (PD-L1) and efficacy.

DETAILED DESCRIPTION:
Dose escalation study: Primary purpose: To investigate the safety and tolerability of GLS-010 in subjects with advanced solid tumors (mainly gastric cancer, esophageal cancer). Secondary purpose: 1. To characterize the pharmacokinetics(PK) profile of GLS-010; 2. To determine dose-limiting toxicity(DLT), maximum tolerated dose (MTD) and recommended Phase II dose (RP2D) for GLS-010; 3. To assess the preliminary anti tumor activity of GLS-010; 4. To assess programmed cell death-1 (PD-1) receptor occupancy. Exploratory purpose: 1. To investigate the preliminary relationship between the expression of the ligand of PD-1 (PD-L1) /PD-L2 and efficacy; 2. To characterize immunogenicity of GLS-010. Expansion study: Primary purpose: To assess the preliminary anti-tumor activity of GLS-010 in subjects with advanced solid tumors(gastric cancer, esophageal cancer); Secondary purpose: 1. To further assess the safety and tolerability of GLS-010; 2. To further assess the safety and tolerability of GLS-010 in subjects with advanced tumors. Exploratory purpose: 1. To assess PD-1 receptor occupancy of GLS-010; 2. To assess the relationship between the expression of PD-L1/PD-L2 and efficacy; 3. To further assess the immunogenicity of GLS-010.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the clinical trial. Provide written informed consent prior to any study-specific screening procedures. Willingness and capability to comply with the requirements of the study;
* Male or female, Age between 18 and 75 years old (margin included) on the day of signing informed consent.
* Imaging and histologically/cytologically confirmed diagnosis of advanced solid tumor;Dose escalation study: Subjects with advanced solid tumor (mainly gastric cancer, esophageal cancer)Expansion study: It is estimated that subjects with gastric cancer and esophageal cancer are to be enrolled. The specific cancer type is to be identified later regarding the dose escalation study result.
* Paraffin embedding sample or biopsy sample available during screening, or be willing to provide tissue from a newly obtained core or excisional biopsy.
* Have no effective standard treatment or are not respond to standard treatment.
* Must have at least one measurable lesion as defined per RECIST Version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Has a predicted survival period ≥ 12 weeks.
* Demonstrate adequate organ and hematopoietic function as defined below. a) Hemoglobin (HGB)≥90 g/L;b)White blood cell count (WBC) ≥3×109/L;c)Absolute neutrophil count (ANC) ≥1.5×109/L;d)Platelets ≥100×109/L;e) Serum total bilirubin (TBIL) ≤ 1.5 X upper limit of normal ULN;f) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 X ULN or ≤5 X ULN for subjects with liver metastases;g)Serum creatinine ≤1.5 X ULN;h)International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN.
* Since signing the ICF, female or male subjects of childbearing potential should be willing to use an adequate method of contraception with the spouse for the course of the study through 5 months after the last dose of study medication

Exclusion Criteria:

* Subjects with meningeal or symptomatic central nervous system metastases.
* Patients with any autoimmune disease, i.e., but not limited to, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (hypothyroidism without clinical symptoms or caused by radiotherapy and chemotherapy can be included); Patients with vitiligo or asthma CR in Childhood, not requiring any intervention in adulthood are permitted to enroll.; patients with asthma requiring a bronchiectasis intervention are not permitted to enroll.
* Subjects who require systemic corticosteroids (at doses equivalent to or greater than 10 mg/day of prednisone) or other immunosuppressive drugs within 14 days prior to or during the study.
* Subjects who have received anti-tumor vaccine or who have received anti-tumor drug treatment with immune-stimulating effect within 4 weeks prior to screening.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti CTLA-4 antibody (including Ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Presence of other active cancers within 5 years prior to enrollment. Patients with cervical carcinoma in situ/ cured skin basal cell carcinoma who have received definitive adequate treatment are eligible.
* Participants with active viral hepatitis (positive HepB sAg and/or positive HepB core Ab with positive HepB DNA>103 copies/mL, or positive HepC antibody), or syphilis positive.
* Subjects with a history of infection with human immunodeficiency virus, or other acquired, congenital immunodeficiency disease, or organ transplantation.
* Subjects with active tuberculosis infection or active tuberculosis infection within 1 year prior to administration, or subjects with active tuberculosis infection more than 1 year prior to administration without formal treatment.
* Subjects with active infection or unexplained fever >38.5℃ during screening and prior to first administration (subject with fever caused by tumor may be included in the group as determined by the investigator).
* History of allergic reactions attributed to any macromolecular protein preparation/monoclonal antibody, or any other composition of the study drug.
* Investigational drug therapy outside of this trial during or within 4 weeks prior to administration.
* Has had prior chemotherapy, radiation therapy, targeted small molecule therapy or major surgery within 2 weeks prior to administration; who has not recovered (i.e. ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent (alopecia excluded)
* Poorly controlled heart disease, such as uncontrolled hyper hypertension, unstable angina pectoris, myocardial infarction within 6 months prior to screening, arrhythmias(including male QTc intervals≥ 450 ms, female QTc intervals≥ 470 ms, QTc intervals calculated by Formula Fridericia).
* Has history of Interstitial Lung Disease or non-infectious pneumonitis. (Patients caused by radiotherapy are eligible)
* Has history of alcoholism or drug abuse within 1 year.
* Has clear history of neurological or mental disorders, i.e. epilepsy, dementia, and poor compliance.
* Other conditions that do not permit compliance with the protocol, evaluated by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of GLS-010 by assessing the percentage of participants who experience a dose-limiting toxicity (DLT) | 28 days after patient enrolled
  To investigate the safety and tolerance profile tolerance profile and the preliminary anti-tumor activity of GLS-010 in subjects with advanced solid tumors ( gastric cancer, esophageal cancer)

SECONDARY OUTCOMES:
Dose Escalation: Area under the plasma concentration time curve (AUC) of GLS-010 | within 2 years after patient enrolled
  To characterize the pharmacokinetics(PK) profile of GLS-010
severity, seriousness, and relatedness of adverse events | within 2 years of last patient enrolled
  Descriptive statistics will be used to summarize results
Dose Escalation: Maximum concentration (Cmax) of GLS-010 | within 2 years after patient enrolled
  To characterize the pharmacokinetics(PK) profile of GLS-010
Dose Escalation: Half life Period (t1/2) of GLS-010 | within 2 years after patient enrolled
  To characterize the Ppharmacokinetics(K) profile of GLS-010

OTHER OUTCOMES:
The percent of PD-1 receptor occupancy | within 2 years of last patient enrolled
  To assess PD-1 receptor occupancy of GLS-010

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MM, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu D, Ma C, Lu P, Gong J, Ye D, Wang S, Peng P, Bai Y, Song Y, Chen J, Jiang O, Zhang G, Ba Y, Chen L, Pan J, Li Q, Zhang L, Gu S, Yin X, Cao B, Han W, Dong H, Guo J, Zhang H, Su H, Jiang Y, Ouyang W, Ma L, Sun Y, Zhang F, Lv J, Guo Y, Xu C, Qi J, Wang L, Wang X, Liu Z, Shen L. Dose escalation and expansion (phase Ia/Ib) study of GLS-010, a recombinant fully human antiprogrammed death-1 monoclonal antibody for advanced solid tumors or lymphoma. Eur J Cancer. 2021 May;148:1-13. doi: 10.1016/j.ejca.2021.01.020. Epub 2021 Mar 7. PMID 33691262